CLINICAL TRIAL: NCT02795377
Title: Hypertension, Endothelial Microparticle Release, and Endothelial Function: Role of Pressure, Shear, and Stretch
Brief Title: Hypertension and Injury
Status: Completed | Type: Observational
Sponsor: Klinik für Kardiologie, Pneumologie und Angiologie (Other)
Responsible Party: Sponsor-Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Principal Investigaor, Heinrich-Heine University, Duesseldorf
Organization: Heinrich-Heine University, Duesseldorf (Other)
Other Study IDs: Hypertension and Injury; 12-011 (Other: CTSU)
Record Dates: First submitted 2016-05-11; First posted 2016-06-10 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Arterial Hypertension; CAD
Keywords: arterial hypertension; microparticle; endothelial function
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- male subjects with arterial hypertension: Measurements will be taken at baseline.
- male subjects without arterial hypertension and no CAD: Measurements will be taken at baseline.
- male subjects with hypertensive crises: Measurements will be taken before and after 4 hours and normalization of arterial blood pressure by urapidil.
- male subjects with stable CAD: Measurements will be taken before and after transfemoral coronary diagnostic angiography.

SUMMARY:
Membrane microparticles are submicron fragments of membrane vesicles shed from various cell types. Circulating endothelial microparticles have been proposed as markers of endothelial injury. However, which mechanical forces contribute to their release is not clear.

DETAILED DESCRIPTION:
In a first series subjects (50% hypertensives) with and without arterial hypertension and no Coronary Artery Disease (CAD) (n=50) will be recruited. MP subpopulations will be discriminated by flow cytometry according to the expression of established surface antigens including CD31+/41-, CD144+, and CD62e+. Besides office and ambulatory 24h blood pressure measurements, pulse wave analysis will be performed to determine central blood pressure, augmentation index (AIX), and pulse wave velocity. Endothelial function (Flow-mediated dilation, FMD), arterial pulsatile stretch (fractional diameter changes, FDC), and wall-shear-stress (WSS) will be measured in the same segment of the brachial artery (BA) by ultrasound. In a second series, the investigators will take measurements in subjects with hypertensive crises (SBP>180 mmHg) (n=20) before and after 4h and normalization of arterial BP by urapidil. In a third series, the investigators will take measurement in subjects with stable CAD (n=10) before and after transfemoral coronary diagnostic angiography.

ELIGIBILITY:
Inclusion Criteria:

* male subjects with or without arterial hypertension, hypertensive crises, stable CAD
* written informed consent

Exclusion Criteria:

* subjects with manifest peripheral artery, or cerebrovascular disease, acute inflammation (CRP>0.6 mg/dl), malignancies, arrhythmias

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with or without arterial hypertension
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-04; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
endothelial function | Baseline
  endothelial function measured by flow-mediated dilation (FMD) for Subgroup 1 and 2
Changes in endothelial function | Baseline and after 4 hours
  endothelial function measured by flow-mediated dilation (FMD) for Subgroup 3
Changes in endothelial function | Baseline and 4 hours after procedure
  endothelial function measured by flow-mediated dilation (FMD) for Subgroup 4 before and after transfemoral coronary diagnostic angiography

SECONDARY OUTCOMES:
Microparticle | Baseline
  Microparticles (CD31+/41-, CD144+, and CD62e+) will be discriminated by flow cytometry for Subgroup 1 and 2
Changes in Microparticle | Baseline and after 4 hours
  Microparticles (CD31+/41-, CD144+, and CD62e+) will be discriminated by flow cytometry for Subgroup 3
Changes Microparticle | Baseline and 4 hours after procedure
  Microparticles (CD31+/41-, CD144+, and CD62e+) will be discriminated by flow cytometry for Subgroup 4 before and after transfemoral coronary diagnostic angiography
Wall Shear Stress | Baseline
  measured by ultrasound in brachial artery for Subgroup 1 and 2
Changes in Wall Shear Stress | Baseline and 4 hours
  measured by ultrasound in brachial artery for Subgroup 3
Changes in Wall Shear Stress | Baseline and 4 hours after procedure
  measured by ultrasound in brachial artery for Subgroup 4 before and after transfemoral coronary diagnostic angiography
changes in fractional diameter (FDC) | Baseline
  measured by ultrasound in brachial artery for Subgroup 1 and 2
changes in fractional diameter (FDC) | Baseline and after 4 hours
  measured by ultrasound in brachial artery for Subgroup 3
Changes in fractional diameter (FDC) | Baseline and 4 hours after procedure
  measured by ultrasound in brachial artery for Subgroup 4 before and after transfemoral coronary diagnostic angiography
pulse wave velocity | Baseline
  measured for Subgroup 1 and 2
Changes in pulse wave velocity | Baseline and after 4 hours
  measured for Subgroup 3
Changes in pulse wave velocity | Baseline and 4 hours after procedure
  measured for Subgroup 4 before and after transfemoral coronary diagnostic angiography
augmentation index | baseline
  measured for Subgroup 1 and 2
Changes in augmentation index | Baseline and after 4 hours
  measured for Subgroup 3
Changes in augmentation index | Baseline and 4 hours after procedure
  measured for Subgroup 4 before and after transfemoral coronary diagnostic angiography

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Sansone, MD, Principal Investigator — Division of Cardiology, Pulmonary Disease and Vascular Medicine
Locations (1):
- Division of Cardiology, Pulmonology and Vascular Medicine Duesseldorf,, Düsseldorf, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Sansone R, Baaken M, Horn P, Schuler D, Westenfeld R, Amabile N, Kelm M, Heiss C. Release of endothelial microparticles in patients with arterial hypertension, hypertensive emergencies and catheter-related injury. Atherosclerosis. 2018 Jun;273:67-74. doi: 10.1016/j.atherosclerosis.2018.04.012. Epub 2018 Apr 12. PMID 29684662